CLINICAL TRIAL: NCT07302477
Title: Growth and Feeding Tolerance of Infants Consuming a Formula Supplemented With Human Milk Oligosaccharides (HMOs): An Uncontrolled, Open-label, Prospective Study
Brief Title: Human Milk Oligosaccharides (HMOs) - Post Marketing Study on Infants (NeHMO)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18.06.INF-Pakistan-TmpDel
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Growth; Tolerance; Adverse Event

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Infants Fed Infant Formula (Experimental): Infant either Fed Exclusive Infant Formula or on Mixed feeding.
  Interventions: Other: HMO Supplemented Infant Formula

INTERVENTIONS:
Other: HMO Supplemented Infant Formula — Starter Infant formula supplemented with 0.18 g /100g powder of 2'FL HMOs,1.2 g protein/100 ml (70% whey) and. B. Lactis.

SUMMARY:
Human milk oligosaccharides (HMOs) represent the third largest solid component of breast milk. Technology advancements made it possible to supplement infant formulas with HMOs (2'FL, LNnT). Two published RCTs have demonstrated that infant formulas supplemented with 2'FL or 2'FL+LNnT are safe, well-tolerated, support normal grow, and may support healthy GI function and confer immune benefits. The performance of HMOs-supplemented formulas assessed in a real-world setting is complementary to previously conducted RCTs conducted in highly controlled clinical settings. Main objectives will be to document the growth and feeding tolerance of healthy term infants consuming an infant formula supplemented with HMOs in a real-world setting. In addition to it considering the potential health/immune benefits of HMOs, it is also important explore the incidences of illnesses (i.e., respiratory illnesses, GI illnesses, and fever) associated with consuming HMOs-supplemented formulas.

DETAILED DESCRIPTION:
Objectives:

The main objective of this study is to document the growth and feeding tolerance of healthy term infants consuming an infant formula supplemented with HMOs for 8 weeks (56 days), in a real-world setting.

Main endpoints:

1. Growth documented via monitoring the anthropometric parameters including weight, length, head circumference, BMI and their corresponding z-scores (i.e., z-scores for weight-for-age, length-for-age, weight-for-length, head circumference-for-age, and BMI-for-age) calculated using the 2006 WHO Growth Standards
2. Feeding tolerance assessed via monitoring parent-reported overall GI symptom burden measured by the Infant Gastrointestinal Symptom Questionnaire (IGSQ) index score (13-item summary score)

Additional objectives:

To describe the following outcomes in infants fed an infant formula supplemented with HMOs:

1. Formula acceptability
2. Despite there are no expected safety concerns, standard Adverse Events (AEs) monitoring will be implemented during the study

Additional endpoints:

1. Formula acceptability assessed by the Study Formula Satisfaction Questionnaire
2. Reported AEs and Serious Adverse Events (SAEs) including type, incidence, severity, seriousness and relation to study formula consumption as well as concomitant medications and non-pharmacological treatments.

   * Select morbidities of interest (i.e., respiratory illnesses, GI illnesses, and fever) will be collected as part of AE reporting and specific corresponding AE guidance forms will be used to standardize reporting of such AEs

Trial design:

Uncontrolled, single arm, open-label, prospective study in infants (enrolled at postnatal age 7 days to 2 months) fed the study formula for 8 weeks (56 days)

Trial population:

Healthy, male and female, term infants, 7 days postnatal age to 2 months of age at the enrollment

Treatment duration:

Total study participation/intervention up to approximately 8 weeks

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of personally signed and dated informed consent document indicating that the infant's parent(s) has been informed of all pertinent aspects of the study
2. Parent(s) Are willing and able to fulfill the requirements of the study protocol
3. Healthy full term (37-42 weeks gestation) infant
4. Be between post-natal age (Date of Birth = Day 0) 7 days to 2 months
5. Parent(s) must have independently elected, before enrollment, to formula feed. IF or mixed feeding. Prior to enrollment parents were counselled about the superiority and advantages of exclusive breastfeeding.

Exclusion Criteria:

1. Had any known case of intolerance/allergy to cow's milk (for formula-fed group only)
2. Had conditions requiring infant feedings other than those specified in the protocol
3. Evidence of significant cardiac, respiratory, endocrinologist, hematologic, gastrointestinal, or other systemic diseases/disorders
4. Parent(s) refusal to participate in the study
5. Infant had consumed any other infant formula in 3 days prior to study start

Ages: 7 Days to 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 125 (Actual)
Dates: Start 2021-07-29 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
World Health Organization (WHO) based weight-for-age z-scores Weight-for-age z-scores using WHO growth standards [Time Frame: 8 weeks (study end)] | 8 Weeks (Study End)
  Weight-for-age z-scores using WHO growth standards
World Health Organization (WHO) based length-for-age z-scores | 8 Weeks (Study End)
  Length-for-age z-scores using WHO growth standards
World Health Organization (WHO) based weight-for-age z-scores | 8 Weeks (Study End)
  Weight-for-length z-scores using WHO growth standards
World Health Organization (WHO) based weight-for-age z-scores | 8 Weeks (Study End)
  head-circumference-for-age z-scores using WHO growth standards
World Health Organization (WHO) based weight-for-age z-scores | 8 Weeks (Study End)
  Weight and height will be combined to calculate BMI in kg/m^2, then BMI-for-age z-scores will be derived using WHO growth standards
Feeding Tolerance | 4 Weeks (Midpoint) and 8 Weeks (Study End Point)
  The Infant Gastrointestinal Symptom Questionnaire (IGSQ) index score will be used to assess GI distress. This is a validated 13-item questionnaire where each item is scored on a scale of 1 to 5 with higher values indicating greater GI distress. A composite IGSQ score is derived from summing the individual scores with a possible range of 13 to 65 where higher values indicate greater GI distress and values ≤23 indicate no digestive distress.

SECONDARY OUTCOMES:
Formula acceptability | 4 Weeks (study midpoint) and 8 weeks (study end point)
  Study Formula Satisfaction Questionnaire
Standard adverse events (AEs) reporting for safety assessment | Time Frame: From the time the informed consent form has been signed at enrollment infant age less than 7 days to 2 months through the 8 weeks of interventio
  Reported adverse events (AEs) and Serious Adverse Events (SAEs) include type, incidence, severity, seriousness and relation to feeding

CONTACTS AND LOCATIONS:
Overall Officials: Huma Fahim, Study Director — Nestle
Locations (4):
- Pakistan (4):
  - Quaid E Azam Medical College, Chak Four Hundred Fifty-four
  - Liaqat National Hospital, Karachi
  - Fatima Memorial Hospital, Lahore
  - Khawaja Muhammad Safdar Medical College, Sialkot

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Storm HM, Shepard J, Czerkies LM, Kineman B, Cohen SS, Reichert H, Carvalho R. 2'-Fucosyllactose Is Well Tolerated in a 100% Whey, Partially Hydrolyzed Infant Formula With Bifidobacterium lactis: A Randomized Controlled Trial. Glob Pediatr Health. 2019 Mar 15;6:2333794X19833995. doi: 10.1177/2333794X19833995. eCollection 2019. PMID 30906817
- See also: 2'-Fucosyllactose Is Well Tolerated in a 100% Whey, Partially Hydrolyzed Infant Formula With Bifidobacterium lactis: A Randomized Controlled Trial — https://pubmed.ncbi.nlm.nih.gov/30906817/